CLINICAL TRIAL: NCT02176460
Title: A Randomized Controlled Trial of Colchicine for Symptom and Inflammation Modification in Knee Osteoarthritis
Brief Title: Colchicine for Symptom and Inflammation in Knee Osteoarthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke University (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COL-01
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Double-blind; placebo-controlled; randomized; colchicine
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- colchicine (Experimental): 0.5mg twice daily for 16 weeks
  Interventions: Drug: Colchicine
- placebo tablet (Placebo Comparator): 1 tablet twice daily for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — 0.5mg twice daily for 16 weeks
  Other Names: generic colchicine tablets (SIN 12490P)
  Arms: colchicine
Drug: Placebo — 1 tablet twice daily
  Other Names: placebo tablet
  Arms: placebo tablet

SUMMARY:
Uric acid may be involved in the activation of the innate immune response in osteoarthritis (OA) pathology and progression. This suggests that traditional gout therapy may be beneficial for OA. Our goal therefore is to assess colchicine, an existing commercially available agent for gout, for a new therapeutic indication-knee OA. The investigators propose a randomized clinical trial (RCT) of 16 weeks' therapy with standard daily dose oral colchicine or placebo for knee OA. The investigators hypothesize that colchicine will block inflammasome mediated inflammation, thereby improve the signs and symptoms of OA, and reduce synovial fluid, serum and urine inflammatory and biochemical joint degradation biomarkers. This trial will potentially provide data to support a new treatment option for knee OA.

DETAILED DESCRIPTION:
In a knee OA cohort with no clinical evidence or self-report of gout, The investigators recently found a significant correlation of synovial fluid uric acid with radiographic and scintigraphic measures of OA severity [1]. The investigators also observed strong correlations of OA severity (radiographically and scintigraphically determined) and synovial fluid uric acid with synovial fluid Interleukin (IL)-18 and IL-1β; these two cytokines are classically produced during gout attacks by innate immune system activation mediated by uric acid crystal-induced inflammasome assembly in macrophages. These results strongly support the involvement of uric acid and the innate immune system in OA pathology and progression. Whereas in gout flares, uric acid in a crystal form is what triggers the innate immune response, we suspect that in OA, uric acid in a microcrystalline or particulate form is the pathogenic agent -- able to trigger an innate immune response; this leads to release of inflammatory cytokines like IL-18, IL-1β and subsequently tumor necrosis factor - α which perpetuates further cartilage degradation. This new conception of the pathogenesis of OA has very important treatment implications; it suggests that existing therapies for gout may be of benefit in OA. Colchicine may be an effective treatment for OA due to its capacity in suppressing the innate immune response at various levels. At micromolar concentrations colchicine suppresses activation of the crystal-induced (NACHT), (LRR) and (PYD) domains containing protein-3 (NALP3) inflammasome; IL-1β processing and release; and L-selectin expression on neutrophils [2]. At nanomolar concentrations colchicine has blocks the release of a crystal-derived chemotactic factor from neutrophil lysosomes; it blocks neutrophil adhesion to endothelium by modulating the distribution of adhesion molecules on the endothelial cells; and it inhibits urate crystal-induced production of superoxide anions from neutrophils and macrophages. The pain and symptom relieving effects of colchicine for knee OA have been demonstrated in three small but well-performed human randomized controlled trials [3-5]; however, the mechanism of action of colchicine in OA has never been evaluated.

The investigators therefore propose a RCT of colchicine to examine the effects on signs and symptoms of knee OA and to evaluate the mechanism of action through analysis of synovial fluid and systemic biomarker profiles.

Hypothesis: The investigators hypothesize that colchicine will block inflammasome mediated inflammation, thereby improve the signs and symptoms of OA, and reduce synovial fluid serum and urine inflammatory and biochemical joint degradation biomarkers.

Aim 1. To determine whether daily oral colchicine at standard clinical doses (0.5 mg two times daily), compared to placebo, can decrease the pain of symptomatic OA knee and improve function when used as adjunctive daily therapy in addition to background therapy with the patient's current stable analgesic regimen.

Aim 2. To evaluate the mechanism of action of colchicine for reducing knee OA signs and symptoms through analyses of synovial fluid, serum, and urine biomarker profiles - these will interrogate and characterize the state of activation of joint metabolism (joint degradation and synthesis markers), inflammatory mediators, the innate immune system and the NALP3 inflammasome components specifically both before (at baseline) and after 16 weeks therapy (at study end) with oral colchicine versus placebo treatment.

This pilot phase II study uses a double-blinded, randomized, placebo, controlled design. Patients with symptomatic and radiographic knee OA (n=120) will be randomized to colchicine (SIN 12490P) 0.5 mg bid (n=60) or placebo (n=60) daily for 16 weeks. Patients will be permitted to remain on their baseline adjunctive therapy, including non-steroidal anti-inflammatory drugs (NSAIDs) without changes for the duration of the study. They will also be allowed the use of paracetamol not more than 2 g/day as rescue analgesia and pill counting at the end of the study will be conducted to determine the amount of rescue medicine utilized over the course of the 16-week study.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee OA meeting American College of Rheumatology (ACR) criteria
* Radiographic criteria for knee OA with Kellgren-Lawrence (KL) stage of ≥ 2 in at least one knee
* Response positive to the question "do you have pain, aching or stiffness of the knee on most days of the past month
* Score of ≥ 40 out of 100 on a visual analogue scale (VAS) for pain
* Age ≥ 21 years or above
* Male and female subjects and all ethnicities included
* Patients to agree to avoid consuming grapefruit and grapefruit juice while using colchicine
* Ability to provide informed consent

Exclusion Criteria:

* Exposure to a corticosteroid (either parenteral or oral) within 3 months prior to the study enrolment
* Knee arthroscopic surgery within 6 months prior to the study enrolment
* Known history of avascular necrosis, inflammatory arthritis (e.g. Rheumatoid Arthritis), Paget's disease, joint infection, periarticular fracture, neuropathic arthropathy, Reiter's syndrome, or gout involving the knee
* Contraindication to arthrocentesis (warfarin use, bleeding disorder, skin rash or skin infection of signal knee)
* Knee joint replacement;
* History of podagra, active gout or treatment for gout
* Pregnancy or lactation - women of childbearing potential will have serum pregnancy testing (ßHCG) at time of entry prior to any imaging studies (X-ray or MRI); female subjects of childbearing potential must agree to use some form of contraception during the 16 week trial and for 1 week after the end of the trial (over 6 half-life equivalents)
* Renal failure with serum creatinine > 150mmol/L (1.7 mg/dL);
* Hepatic impairment defined by serum alanine transaminase (ALT) above the upper limit of normal for the clinical laboratory performing the screening test
* Muscle impairment defined by elevated serum creatine phosphokinase (CPK) above the upper limit of normal for the clinical laboratory performing the screening test
* Personnel directly affiliated with this study or their immediate family members (defined as a spouse, parent, child or sibling, whether biological or legally adopted)
* Current enrolment in or discontinued within the last 30 days from a clinical trial involving an off-label use of an investigational drug or device, or are concurrently enrolled in any other type of medical research judged to be scientifically or medically incompatible with this study
* Inability to understand and cooperate with the investigators or to give valid consent;
* Contraindication for magnetic resonance imaging (MRI) - this is exclusion only for the subset of individuals selected for this imaging procedure;
* Anticipation of need for joint replacement within 4 months of the start of the intervention;
* Current treatment with drugs known to inhibit Cytochrome 450(3A4) isoforms and/or P-glycoprotein (P-gp) that increase the risk of colchicine-induced toxic effects (see: http://www.fda.gov/Drugs/Drug-safety/PostmarketDrugSafetyInformationforPatientsandProviders/DrugSafetyInformationforHeathcareProfessionals/ucm174315.htm).

Inclusion can be considered after 14 day wash out of agents listed in the drug information sheet, but only if treatment in the near future with one of these agents is not anticipated. The clinical necessity for such treatments during the study will require immediate discontinuation of the study drug and conversion of the patient to standard care. However, the patient will remain on study and scheduled measurements taken. Analyses will be performed on an intention-to-treat basis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
30% improvement in total Western Ontario and McMaster Universities Arthritis Index (WOMAC) of the signal knee. | baseline and week 16
  The primary end point will be 30% improvement in total Western Ontario and McMaster Universities Arthritis Index (WOMAC) of the signal knee.

SECONDARY OUTCOMES:
change in WOMAC pain score and physical function score | baseline and week 16
change in Health Assessment Questionnaire (HAQ) | baseline and week 16
change in quality of life | baseline and week 16
  Medical Outcome Short form 36
quantify of rescue medication used | baseline and week 16
  paracetamol
Change in Synovitis and cartilage morphology on Magnetic Resonance Imaging | baseline and week 16
  In a subgroup of participants (10 participants in interventional arm and 10 participants in placebo arm)
change in synovial fluid Interleukin-18, Interleukin-1β, or tumor necrosis factor -α | baseline and week 16
specific adverse event | from baseline to week 16
  signs or symptoms of colchicine toxicity such as muscle weakness or pain, numbness or tingling in the fingers or toes, diarrhoea, vomiting, elevation of muscle enzyme
OMERACT-ORSI response criteria | week 16
  Outcome Measure in Rheumatology (OMERACT-) - Osteoarthritis Research Society International (ORSI-) response criteria

OTHER OUTCOMES:
Other exploratory outcomes include treatment response of the other biomarker variables. | baseline and week 16
  serum (s)/ synovial fluid (sf) uric acid; inflammasome associated - s/sf IL-1ß, IL-18, tumor necrosis factor α, caspase-1, Toll like receptor (TLR)-2, and TLR-4; oxidant stress - s/sf xanthine oxidase, allantoin, inorganic pyrophosphate and sf carbonyl content; other inflammatory markers - s Cluster of Differentiation 163 (potentially indicative of macrophage activation), s/sf matrix metalloproteinase (MMP)3, IL-6, and high sensitivity C-reactive protein; cartilage degradation markers - sf glycosaminoglycan fragments and sf C-terminal crosslinked telopeptide type II collagen.
Colchicine pharmacogenetics: Cytochrome P450 (CYP3A4) and (CYP3A5) polymorphism | baseline
pharmacokinetics: Peak Plasma Concentration (Cmax) of colchicine | baseline, week 1, week 4 and week 16

CONTACTS AND LOCATIONS:
Overall Officials: Ying Y Leung, MBChB, Principal Investigator — Singapore General Hospital; Virginia Kraus, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leung YY, Haaland B, Huebner JL, Wong SBS, Tjai M, Wang C, Chowbay B, Thumboo J, Chakraborty B, Tan MH, Kraus VB. Colchicine lack of effectiveness in symptom and inflammation modification in knee osteoarthritis (COLKOA): a randomized controlled trial. Osteoarthritis Cartilage. 2018 May;26(5):631-640. doi: 10.1016/j.joca.2018.01.026. Epub 2018 Feb 7. PMID 29426008
- [Derived] Leung YY, Thumboo J, Wong BS, Haaland B, Chowbay B, Chakraborty B, Tan MH, Kraus VB. Colchicine effectiveness in symptom and inflammation modification in knee osteoarthritis (COLKOA): study protocol for a randomized controlled trial. Trials. 2015 Apr 30;16:200. doi: 10.1186/s13063-015-0726-x. PMID 25925674